CLINICAL TRIAL: NCT05801744
Title: Operant Conditioning of Reflex Pathways to Improve Walking in Individuals Post-stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1656292
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Post-stroke Hemiparesis; Foot Drop
MeSH Terms: conditions — Stroke; Peroneal Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reciprocal inhibition up conditioning (Experimental): Each participant completes 6 baseline sessions and 30 up conditioning sessions. In the 30 conditioning sessions, the magnitude of reciprocal inhibition in the paretic leg of participants post-stroke will be up conditioned.
  Interventions: Behavioral: Operant conditioning

INTERVENTIONS:
Behavioral: Operant conditioning — In this training, individuals with post-stroke hemiparesis are trained to increase the amount of reciprocal inhibition in their paretic leg. By increasing the amount of reciprocal inhibition, the paretic ankle in people post-stroke may exhibit less foot drop.

SUMMARY:
The purpose of this study is to examine the changes in reflex pathways in the paretic ankle plantarflexors in individuals with post-stroke hemiparesis using operant conditioning. We are recruiting 5 individuals with chronic post-stroke hemiparesis with foot drop in the affected leg to participate in the reflex training procedure. The study involves 40 visits with a total study duration of about 4 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months following a single, unilateral stroke, resulting in hemiparesis.
* Ambulatory with or without assistive device, but must demonstrate a gait deficit which is indicative of foot drop from reduced activation of the tibialis anterior muscle.
* Able to follow verbal directions.
* Able to see icons on computer monitor (with or without corrective lenses) from at least 4 feet away.
* All subjects will be adults at least 18 years old.
* Know history and current medication management for lower limb spasticity, if any.

Exclusion Criteria:

* No history of ear disease or balance problems outside of those caused by the stroke.
* Cerebellar stroke
* No other neurological disease or injuries other than the stroke affecting the use of the legs and/or walking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in magnitude of reciprocal inhibition | Before training Baseline, after completion of 30 training sessions, and 1 month after the completion of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No